CLINICAL TRIAL: NCT02635152
Title: Evaluation of an Internet-Based Treatment for Body Dysmorphic Disorder
Brief Title: Interpretation Bias Modification for Body Dysmorphic Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Jesse Cougle, Associate Professor, Florida State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017.20244
Record Dates: First submitted 2015-12-16; First posted 2015-12-18 (Estimated); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: Body Dysmorphic Disorder
MeSH Terms: conditions — Body Dysmorphic Disorders | interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpretation Bias Modification (IBM) (Experimental): Treatment consists of eight brief sessions. In Task 1, participants read unique scenarios ("You notice someone pointing in your direction"). A sentence meant to resolve the ambiguity will appear ("This person thinks they reco_nize you"). After filling in the missing letter, the interpretation is reinforced by requiring the participants to correctly answer "yes" or "no" to a comprehension question ("Is this person mocking you?"). In Task 2, participants are shown a word denoting a threatening ("mocking") or benign ("cheerful") interpretation. Participants are presented with an ambiguous scenario ("You hear people at a nearby table laughing") and asked to denote whether the word and the sentence are related. Participants will receive positive or negative feedback based on their response.
  Interventions: Behavioral: Interpretation Bias Modification
- Progressive Muscle Relaxation (PMR) (Active Comparator): Participants will receive eight brief sessions of PMR. They will listen to a PMR script (Kassinove & Tafrate, 2002). Participants will be asked to make sure they are sitting comfortably, close their eyes, and systematically tense and release 10 different muscle groups.
  Interventions: Behavioral: Progressive Muscle Relaxation

INTERVENTIONS:
Behavioral: Interpretation Bias Modification — Eight 10-25 minute sessions of interpretation modification to reduce negative interpretation biases related to appearance.
  Arms: Interpretation Bias Modification (IBM)
Behavioral: Progressive Muscle Relaxation — Eight 15-minute sessions of progressive muscle relaxation (PMR).
  Arms: Progressive Muscle Relaxation (PMR)

SUMMARY:
The purpose of this study is to determine whether a computerized intervention designed to reduce appearance and evaluation related interpretation biases will reduce symptoms associated with body dysmorphic disorder.

DETAILED DESCRIPTION:
The present study aims to examine the feasibility of a remote treatment for body dysmorphic disorder delivered via the Internet. To evaluate the efficacy of the IBM protocol we have developed in reducing negative appearance and evaluative related interpretations, we will conduct a two-arm randomized controlled trial over the internet. Individuals with a diagnosis of body dysmorphic disorder (N = 40) will be randomized to one of two conditions: 1) IBM or 2) progressive muscle relaxation. Each condition will consist of eight 10-25 minute treatment sessions. Participants will complete two sessions per week for four weeks and will be administered assessments at pre-treatment, one week post-treatment and at 3-month follow-up. We hypothesize that: 1) IBM will lead to greater reductions in BDD symptoms than the PMR condition; 2) IBM will lead to greater reductions in depression, anxiety and suicidal ideation than the PMR condition; 3) IBM will lead to greater reductions in threat interpretations and greater increases in benign interpretations than the PMR condition; 4) The effects of condition on BDD symptoms will be mediated by changes in BDD-related interpretation bias; and 5) The effects of training in the IBM condition will be maintained at the 3-month follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

* Current diagnosis of Body Dysmorphic Disorder according to DSM-5 criteria
* BDD-YBOCS score greater than or equal to 20
* Fluent in English
* No significant physical defect or flaw in appearance (e.g., disfiguration)

Exclusion Criteria:

* History of psychotic disorder, bipolar disorder, borderline personality disorder
* Current substance use disorder
* Unstable medication status (i.e. change in medication within the last month)
* Concurrent psychotherapy for appearance concerns
* Active and clinically significant suicidality

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-09; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Scale Modified for Body Dysmorphic Disorder (BDD-YBOCS; Phillips et al., 1997) | change from baseline at one-week post treatment and 3-months post-treatment
  Measures past-week BDD symptom severity

SECONDARY OUTCOMES:
Beck Depression Inventory (BDI-II; Beck, Steer, & Brown, 1996) | change from baseline at one-week post treatment and 3-months post-treatment
  Measures depressive symptom severity
Beck Anxiety Inventory (BAI; Steer & Beck, 1997) | change from baseline at one-week post treatment and 3-months post-treatment
  Measure anxious symptom severity
Depressive Symptom Index-Suicidality Subscale | change from baseline at one-week post treatment and 3-months post-treatment
  Measure severity of recent suicidality
Body Dysmorphic Disorder Word Sentence Association Paradigm (BDD-WSAP; modified from Hindash & Amir, 2011) | change from baseline at one-week post treatment and 3-months post-treatment
  Measure of strength of BDD-related (i.e. evaluation- and appearance- related threat interpretation biases)

CONTACTS AND LOCATIONS:
Overall Officials: Natalie L. Matheny, BA, Principal Investigator — Florida State University
Locations (1):
- Florida State University Psychology Department, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Wilver NL, Cougle JR. An Internet-based controlled trial of interpretation bias modification versus progressive muscle relaxation for body dysmorphic disorder. J Consult Clin Psychol. 2019 Mar;87(3):257-269. doi: 10.1037/ccp0000372. Epub 2018 Dec 27. PMID 30589349